CLINICAL TRIAL: NCT05606744
Title: Effects of Blood Flow Restriction During Multiple-joint Eccentric Resistance Training on Muscle Morphology and Function of the Lower Body
Brief Title: Effects of Blood Flow Restriction During Eccentric Resistance Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Brennan Thompson, Associate Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12042a
Record Dates: First submitted 2022-10-13; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Blood Flow Restriction

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned to a BFR or non BFR exercise condition. The subjects will perform a single, 3-5 minute bout of eccentric exercise on the Eccentron device either with BFR (with restriction cuffs on the thigh per the procedures below) or without the BFR.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric exercise (Active Comparator): Only multi-joint eccentric exercise
  Interventions: Device: Eccentric exercise / Eccentric exercise with blood flow restriction
- Eccentric training with blood flow restriction (Experimental): Multi-joint eccentric exercise with blood flow restriction
  Interventions: Device: Eccentric exercise / Eccentric exercise with blood flow restriction

INTERVENTIONS:
Device: Eccentric exercise / Eccentric exercise with blood flow restriction — Individuals will be randomized to receive eccentric exercise only, or eccentric exercise with blood flow restriction.

SUMMARY:
The purpose of this study is to compare the muscle strength and muscle soreness effects experienced following short term (acute) eccentric exercise with and without blood flow restriction (BFR) performed at low - moderate training intensities.

ELIGIBILITY:
Exclusion Criteria:

* lower body surgery or injury in the last 12 months
* have any neuromuscular disease
* height >76 inches tall
* height <54 inches tall
* eccentric strength greater than 725 pounds
* pregnant or plan to be pregnant in the duration of the protocol
* don't do resistance exercise at least once per week
* perform intense cardio or strength training >4 days per week
* Present with any other significant comorbid conditions that would impair the ability to participate in the exercise-based testing

Inclusion criteria:

* 18 - 30 years old
* strength train lower body 1-3 times per week

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (soreness) | Baseline (pretest)
  soreness
visual analog scale (soreness) | immediately post exercise
  soreness
visual analog scale (soreness) | 24 hours post exercise
  soreness
visual analog scale (soreness) | 48 hours post exercise
  soreness
visual analog scale (soreness) | 72 hours post exercise
  soreness
force algometer (soreness) | Baseline (pretest)
  soreness
force algometer (soreness) | immediately post exercise
  soreness
force algometer (soreness) | 24 hours post exercise
  soreness
force algometer (soreness) | 48 hours post exercise
  soreness
force algometer (soreness) | 72 hours post exercise
  soreness

SECONDARY OUTCOMES:
Eccentric muscle strength | Baseline (pretest)
  muscle strength will be assessed on the Eccentron.
Eccentric muscle strength | immediately post exercise
  muscle strength will be assessed on the Eccentron.
Eccentric muscle strength | 24 hours post exercise
  muscle strength will be assessed on the Eccentron.
Eccentric muscle strength | 48 hours post exercise
  muscle strength will be assessed on the Eccentron.
Eccentric muscle strength | 72 hours post exercise
  muscle strength will be assessed on the Eccentron.
Single-leg hop | Baseline (pretest)
  3 single-leg hops per limb
Single-leg hop | immediately post exercise
  3 single-leg hops per limb
Single-leg hop | 24 hours post exercise
  3 single-leg hops per limb
Single-leg hop | 48 hours post exercise
  3 single-leg hops per limb
Single-leg hop | 72 hours post exercise
  3 single-leg hops per limb

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Thompson, PhD, Principal Investigator — Utah State University

IPD SHARING:
Plan to Share IPD: Undecided